CLINICAL TRIAL: NCT02576574
Title: A Phase III, Open-label, Multicenter Trial of Avelumab (MSB0010718C) Versus Platinum-based Doublet as a First-line Treatment of Recurrent or Stage IV PD-L1+NSCLC
Brief Title: Avelumab in First-line NSCLC (JAVELIN Lung 100)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 100070-005; 2015-001537-24 (EudraCT Number)
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Results first posted 2023-01-04 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: First Line Non-Small Cell Lung Cancer
Keywords: Avelumab; MSB0010718C; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — avelumab; Pemetrexed; Paclitaxel; Gemcitabine; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Avelumab Biweekly (Experimental)
  Interventions: Drug: Avelumab
- Avelumab Weekly (Experimental)
  Interventions: Drug: Cisplatin; Drug: Avelumab Weekly
- Chemotherapy (Active Comparator)
  Interventions: Drug: Pemetrexed; Drug: Paclitaxel; Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Avelumab — Participants received Avelumab at a dose of 10 milligrams per kilogram (mg/kg) as a 1-hour (-10/+20 minutes) intravenous (IV) infusion once every 2 weeks until disease progression or unacceptable toxicities.
  Other Names: Anti-PD-L1; MSB0010718C
  Arms: Avelumab Biweekly
Drug: Pemetrexed — Participants received Pemetrexed 500 milligrams per square meter (mg/m^2) by IV infusion on Day 1 of 3-Week cycle up to a maximum of 6 cycles of IV injection until disease progression or unacceptable toxicities.
  Arms: Chemotherapy
Drug: Paclitaxel — Participants received Paclitaxel 200 mg/m^2 by IV infusion on Day 1 of 3-Week cycle up to a maximum of 6 cycles of IV injection until disease progression or unacceptable toxicities.
  Arms: Chemotherapy
Drug: Gemcitabine — Participants received Gemcitabine 1250 mg/m^2 on Day 1 and Day 8 by IV infusion in 3-Week cycle up to a maximum of 6 cycles when combined with cisplatin of IV injection until disease progression or unacceptable toxicities.
  Arms: Chemotherapy
Drug: Gemcitabine — Participants received Gemcitabine 1000 mg/m^2 on Day 1 and Day 8 by IV infusion in 3-Week cycle up to a maximum of 6 cycles of IV injection when combined with carboplatin until disease progression or unacceptable toxicities.
  Arms: Chemotherapy
Drug: Carboplatin — Participants received Carboplatin area under concentration curve (AUC) 5 mg/mL*min in 3-Week cycle up to a maximum of 6 cycles of IV injection when combined with gemcitabine until disease progression or unacceptable toxicities.
  Arms: Chemotherapy
Drug: Cisplatin — Participants received Cisplatin 75 mg/m^2 by IV infusion in 3-Week cycle up to a maximum of 6 cycles of IV injection until disease progression or unacceptable toxicities.
  Arms: Avelumab Weekly
Drug: Carboplatin — Carboplatin AUC 6 mg/mL*min by IV infusion in 3-Week cycle up to a maximum of 6 cycles of IV injection when combined with pemetrexed, or paclitaxel until disease progression or unacceptable toxicities.
  Arms: Chemotherapy
Drug: Avelumab Weekly — Participants received Avelumab at a dose of 10 mg/kg as a 1-hour (-10/+20 minutes) IV infusion every week for 12 consecutive weeks.
  Other Names: Anti-PD-L1; MSB0010718C
  Arms: Avelumab Weekly

SUMMARY:
The purpose of this study was to demonstrate superiority with regard to Overall Survival (OS) or Progression Free Survival (PFS) of avelumab versus platinum-based doublet, based on an Independent Review Committee assessment, in Non-small cell lung cancer (NSCLC) participants with Programmed death ligand 1+ (PD-L1+) tumors.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged greater than or equal to (>=) 18 years
* With Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1 at trial entry
* At least 1 measurable tumor lesion
* With histologically confirmed metastatic or recurrent (Stage IV) non-small cell lung cancer (NSCLC)
* With availability of a recently-obtained, formalin-fixed, paraffin-embedded (FFPE) tissue sample containing tumor (biopsy from a non-irradiated area preferably within 6 months) or a minimum number of 10 (preferably 25) unstained tumor slides cut within 1 week, and suitable for PD-L1 expression assessment
* Subjects must not have received any treatment for systemic lung cancer, and have an estimated life expectancy of more than 12 weeks
* Other protocol defined criteria could apply

Exclusion Criteria:

* Subjects whose disease harbors a EGFR mutation, or anaplastic lymphoma kinase (ALK) rearrangement are not eligible.
* Other exclusion criteria include prior therapy with any antibody or drug targeting T cell coregulatory proteins, concurrent anticancer treatment, or immunosuppressive agents
* Known severe hypersensitivity reactions to monoclonal antibodies (Grade >= 3 NCI CTCAE v 4.03), history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma), and persisting toxicity related to prior therapy of Grade > 1 NCI-CTCAE v 4.03.
* Subjects with brain metastases are excluded, except those meeting the following criteria: brain metastases that have been treated locally and are clinically stable for at least 2 weeks prior to randomization, subjects must be either off steroids or on a stable or decreasing dose of <= 10 mg daily prednisone (or equivalent), and do not have ongoing neurological symptoms that are related to the brain localization of the disease.
* Other protocol defined criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1214 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2024-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., an affiliate of Merck KGaA, Darmstadt, Germany
Locations (348):
- United States (21):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Arizona Center for Cancer Care, Surprise, Arizona
  - Sharp Memorial Hospital, San Diego, California
  - University Cancer Institute, Boynton Beach, Florida
  - South Georgia Medical Center, Valdosta, Georgia
  - Christus Cancer Treatment Center, Shreveport, Louisiana
  - Henry Ford Hospital, Detroit, Michigan
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - San Juan Oncology Associates, Farmington, New Mexico
  - Novant Health Oncology Specialists, Kernersville, North Carolina
  - Mercy Research, Oklahoma City, Oklahoma
  - Kaiser Permanente Northwest, Portland, Oregon
  - Lancaster Cancer Center, Lancaster, Pennsylvania
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - Oncology Consultants, P.A., Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - Cheyenne Regional Medical Center, Cheyenne, Wyoming
- Australia (14):
  - Albury Wodonga Regional Cancer Centre, Albury, New South Wales
  - Coffs Harbour Health Campus, Coffs Harbour, New South Wales
  - St George Private Hospital, Kogarah, New South Wales
  - Lismore Base Hospital, Lismore, New South Wales
  - Orange Health Service, Orange, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Gallipoli Medical Research Foundation Ltd, Greenslopes, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Ballarat Base Hospital, Ballarat, Victoria
  - Bendigo Hospital, Bendigo, Victoria
  - South West Healthcare, Warrnambool, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Belgium (3):
  - ZNA Middelheim, Antwerp
  - A.Z. Klina, Brasschaat
  - CHU Ambroise Paré, Mons
- Brazil (20):
  - CRIO - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - NOB - Núcleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - CEBROM - Centro Brasileiro de Radioterapia, Oncologia e Mastologia, Goiânia, Goiás
  - Hospital Erasto Gaertner - Liga Paranaense de Combate ao Câncer, Curitiba, Paraná
  - Hospital de Caridade de Ijuí, Ijuí, Rio Grande do Sul
  - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - IMV-Pesquisa Cardiologica Sociedade Simples - HMD - COR, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceição, Porto Alegre, Rio Grande do Sul
  - CEPON - Centro de Pesquisas Oncológicas de Santa Catarina, Florianópolis, Santa Catarina
  - Clínica de Neoplasias Litoral Ltda., Itajaí, Santa Catarina
  - Hospital de Câncer de Barretos - Fundação Pio XII, Barretos, São Paulo
  - Fundação Doutor Amaral Carvalho, Jaú, São Paulo
  - CEPHO - Centro de Estudos e Pesquisas em Hematologia e Oncologia, Santo André, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - ICESP - Instituto do Câncer do Estado de São Paulo Octavio Frias de Oliveira, São Paulo, São Paulo
  - IBCC - Instituto Brasileiro de Controle do Câncer, São Paulo, São Paulo
  - INCA - Instituto Nacional de Câncer, Rio de Janeiro
- Bulgaria (4):
  - Complex Oncological Center - Ruse, EODD, Rousse
  - MHAT for women's health - Nadezhda, OOD, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - Shato, Ead, Sofia
- Canada (2):
  - The Moncton Hospital, Moncton, New Brunswick
  - Mount Sinai Hospital, Toronto, Ontario
- Chile (8):
  - FALP - Fundación Arturo López Pérez, Santiago
  - Clinica Santa Maria, Santiago
  - IRAM - Instituto de Radio Medicina, Santiago
  - Hospital Militar de Santiago, Santiago
  - Hospital Clínico San Borja Arriaran, Santiago
  - Hospital Clínico Universidad de Chile, Santiago
  - Hospital Clinico Viña del Mar, Viña del Mar
  - Centro de Investigaciones Clinicas Viña del Mar, Viña del Mar
- China (5):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Linyi Cancer Hospital, Linyi, Shandong
- Colombia (4):
  - Administradora Country S.A., Bogotá
  - Fundación Oftalmológica de Santander - FOSCAL, Floridablanca
  - Hospital Pablo Tobón Uribe, Medellín
  - IPS IMAT- Instituto Medico de Alta Tecnologia - Oncomedica S.A., Montería
- Croatia (2):
  - University Clinic for Pulmonary Diseases, Zagreb
  - University Hospital Centre "Sestre Milosrdnice", Zagreb
- Bank of Cyprus Oncology Center, Nicosia, Cyprus
- Czechia (6):
  - Krajska nemocnice Liberec, a.s., Liberec
  - Nemocnice Na Plesi s.r.o., Nová Ves pod Pleší
  - Fakultni nemocnice Olomouc, Olomouc
  - Vitkovicka nemocnice a.s, Ostrava - Vitkovice
  - Thomayerova nemocnice, Praha 4 - Krc
  - Krajska zdravotni, a.s. - Masarykova nemocnice v Usti nad Labem, o.z., Ústí nad Labem
- Denmark (2):
  - Herning Sygehus, Herning
  - Roskilde Sygehus, Roskilde
- North Estonia Medical Centre Foundation, Tallinn, Estonia
- France (15):
  - Centre Antoine Lacassagne, Nice, Alpes Maritimes
  - CHU de Strasbourg - Nouvel Hôpital Civil, Strasbourg, Bas Rhin
  - Hôpital privé Clairval, Marseille, Bouches-du-Rhône
  - Hôpital Nord - AP-HM Marseille#, Marseille, Bouches-du-Rhône
  - CHU Besançon - Hôpital Jean Minjoz, Besançon, Doubs
  - CHU Brest - Hôpital Morvan, Brest, Finistere
  - Groupe Hospitalier Sud - Hôpital Haut-Lévêque, Pessac, Gironde
  - CHU Angers - Hôpital Hôtel Dieu#, Angers, Maine Et Loire
  - Hôpital Cochin, Paris, Paris
  - Centre Hospitalier de la Côte Basque, Bayonne, Pyrenees Atlantiques
  - Centre Hospitalier de la Croix Rousse, Lyon, Rhone
  - Clinique Victor Hugo - Centre Jean Bernard, Le Mans, Sarthe
  - Institut Sainte Catherine, Avignon, Vaculuse
  - Centre Hospitalier Intercommunal de Créteil, Créteil, Val De Marne
  - Hôpital Saint-Louis - Paris, Paris
- Germany (2):
  - Universitaetsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - LungenClinic Grosshansdorf GmbH, Großhansdorf, Schleswig-Holstein
- Greece (8):
  - 251 General Air Force Hospital, Athens
  - General Hospital of Athens of Chest Diseases "SOTIRIA", Athens
  - University General Hospital "Attikon", Athens
  - General Oncology Hospital of Kifissia " Agioi Anargyroi", Athens
  - Metropolitan General Hospital, Athens
  - University General Hospital of Heraklion, Heraklion
  - University General Hospital of Patra, Pátrai
  - Euromedica General Clinic Thessaloniki, Thessaloniki
- Hungary (10):
  - Orszagos Koranyi Pulmonologiai Intezet, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Semmelweis Egyetem, Budapest
  - Csongrad Megyei Mellkasi Betegsegek Szakkorhaza, Deszk
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Borsod-Abauj-Zemplen Megyei Kozponti Korhaz es Egyetemi Oktatokorhaz, Miskolc
  - SzSzB Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
  - Tudogyogyintezet Torokbalint, Törökbálint
  - Zala Megyei Szent Rafael Korhaz, Zalaegerszeg
- Cork University Hospital, Cork, Ireland
- Israel (9):
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care Center, Haifa
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Sapir Medical Center, Meir Hospital, Kfar Saba
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Assaf Harofeh, Rishon LeZiyyon
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (7):
  - Ospedale Mater Salutis, Legnago, Verona
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia
  - Presidio Ospedaliero Garibaldi Nesima, Catania
  - Azienda Ospedaliero Universitaria San Martino, Genova
  - Seconda Università degli Studi di Napoli, Napoli
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Azienda Ospedaliero Universitaria Pisana, Pisa
- Japan (13):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - NHO Hokkaido Cancer Center, Sapporo, Hokkaido
  - Institute of Biomedical Research and Innovation Hospital, Kobe, Hyōgo
  - Kobe City Hospital Organization Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Yokohama Municipal Citizen's Hospital, Yokohama, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Osaka Medical College Hospital, Takatsuki-shi, Osaka
  - National Cancer Center Hospital, Chūōku, Tokyo-To
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo-To
  - Toyama University Hospital, Toyama, Toyama
  - Kobe City Hospital Organization Kobe City Medical Center General Hospital, Kobe
- Lebanon (5):
  - American University of Beirut Medical Center, Beirut
  - Rafik Hariri University Hospital, Beirut
  - Hotel Dieu de France Hospital, Beirut
  - Mount Lebanon Hospital, Beirut
  - Hammoud Hospital University Medical Center, Saida
- Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas, Lithuania
- Netherlands (3):
  - Martini Ziekenhuis, Groningen
  - Westfriesgasthuis - PARENT, Hoorn
  - ETZ Elisabeth, Tilburg
- New Zealand (6):
  - Auckland City Hospital, Auckland
  - Dunedin Public Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - Palmerston North Hospital, Palmerston North
  - Tauranga Hospital, Tauranga
  - Wellington Hospital, Wellington
- Peru (3):
  - Instituto Nacional de Enfermedades Neoplásicas, Lima
  - Clinica Internacional Sede San Borja, Lima
  - Oncosalud, Lima
- Poland (11):
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska sp. komandytowo-akcyjna, Lodz
  - Instytut MSF Sp. o.o, Lodz
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Łodzi, Lodz
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - SSZZOZ im. Dr Teodora Dunina w Rudce, Mrozy
  - SP Zespol Gruzlicy i Chorob Pluc w Olsztynie, Olsztyn
  - Mazowieckie Centrum Leczenia Chorob Pluc i Gruzlicy, Otwock
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego, Poznan
  - Izerskie Centrum Pulmonologii i Chemioterapii "IZER-MED" Spolka z o.o., Szklarska Poręba
  - Centrum Onkologii-Instytut im. M. Sklodowskiej Curie, Warsaw
  - Mazowiecki Szpital Onkologiczny, Wieliszew
- Portugal (12):
  - Hospital Garcia de Orta, EPE, Almada
  - Hospital Professor Doutor Fernando Fonseca, E.P.E., Amadora-Lisbon
  - Centro Hospitalar De Coimbra-CHUC, Coimbra
  - Centro Hospitalar e Universitário de Coimbra, E.P.E (CHC), Coimbra
  - Centro Hospitalar de Lisboa Norte, E.P.E. - Hospital Pulido Valente, Lisbon
  - Centro Hospitalar de Lisboa Central, E.P.E. - Hospital de Santo António dos Capuchos, Lisbon
  - Centro Hospitalar do Porto, E.P.E. - Hospital de Santo António, Porto
  - Hospital CUF Porto, Porto
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE, Porto
  - Centro Hospitalar de São João, E.P.E., Porto
  - Centro Hospitalar de Entre o Douro e Vouga, E.P.E - Hospital de São Sebastião, Santa Maria da Feira
  - Centro Hospitalar Vila Nova de Gaia/Espinho, E.P.E, Vila Nova de Gaia
- Romania (17):
  - Spitalul Judetean de Urgenta "Dr. Constantin Opris" Baia Mare, Baia Mare
  - S.C Policlinica de Diagnostic Rapid S.A, Brasov
  - Institutul Oncologic "Prof. Dr. Al. Trestioreanu", Bucharest
  - Spitalul Clinic Coltea, Bucharest
  - S.C Gral Medical S.R.L, Bucharest
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta" Cluj Napoca, Cluj-Napoca
  - S.C Medisprof S.R.L, Cluj-Napoca
  - Spitalul Militar de Urgenta "Dr.Constantin Papilian"Cluj -Napoca, Cluj-Napoca
  - S.C Radiotherapy Center Cluj S.R.L, Comuna Floresti
  - Spitalul Clinic Judetean de Urgenta "Sf. Apostol Andrei" Constanta, Constanța
  - S.C Centrul de Oncologie Sf. Nectarie S.R.L, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
  - S.C Pelican Impex S.R.L, Oradea
  - Spitalul Clinic Municipal "Dr. Gavril Curteanu" Oradea, Oradea
  - Spitalul Judetean de Urgenta "Sf. Ioan cel Nou" Suceava, Suceava
  - S.C Oncocenter Oncologie Clinica S.R.L, Timișoara
  - S.C Oncomed S.R.L, Timișoara
- Russia (24):
  - SBIH of Arkhangelsk region "Arkhangelsk Clinical Oncological Dispensary", Arkhangelsk
  - LLC Evimed, Chelyabinsk
  - Chelyabinsk Regional Oncology Dispensary, Chelyabinsk
  - Irkutsk Regional Oncology Dispensary, Irkutsk
  - RBIH "Ivanovo Regional Oncological Dispensary", Ivanovo
  - SBHI of Kaluga Region "Kaluga regional clinical oncology dispensary", Kaluga
  - SAIH "Republican Clinical Oncological Dispensary of the Ministry of Healthcare of Republic Tatarstan, Kazan'
  - Kemerovo SPI Regional Clinical Oncology Dispensary, Kemerovo
  - SBHI "Krasnoyarsk Regional Oncology Dispensary n.a. A.I. Kryzhanovsky", Krasnoyarsk
  - RBIH "Kursk regional clinical oncology dispensary" of Kursk Region Healthcare Committee, Kursk
  - FSBSI "Russian Oncological Scientific Center n.a. N.N. Blokhin", Moscow
  - Murmansk Regional Clinical Hospital named after Bayandin, Murmansk
  - SBHI of Novosibirsk region "Novosibirsk Regional Oncological Dispensary", Novosibirsk
  - SBIH of Stavropol territory "Pyatigorsk Oncological Dispensary", Pyatigorsk
  - FSBHI Clinical research institute of phthisiopulmonology, Saint Petersburg
  - SBIH "Leningrad Regional Oncological Dispensary", Saint Petersburg
  - "Bio Eq" LLC, Saint Petersburg
  - FBI "Scientific Research Institute of Oncology n. a. N. N. Petrov", Saint Petersburg
  - SBIH "Samara Regional Clinical Oncological Dispensary", Samara
  - SBIH "Oncological Dispensary # 2" of the MoH of Krasnodar territory, Sochi
  - Tomsk Research Instutite of Oncology, Tomsk
  - BHI of Omsk region "Clinical Oncology Dispensary", Tomsk
  - Medicinskiy gorod, Tyumen
  - SBIH of Yaroslavl region "Regional Clinical Oncological Hospital", Yaroslavl
- Serbia (7):
  - Clinical Center of Serbia, Belgrade
  - Institute of Oncology and Radiology of Serbia, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center Bezanijska Kosa, Belgrade
  - Clinical Center Nis, Pulmonary Diseases Clinic, Gornji Matejevac
  - Institute for Pulmonary Diseases of Vojvodina, Kamenitz
  - Clinical Center Kragujevac, Kragujevac
- Singapore (3):
  - National University Cancer Institute, Singapore
  - National Cancer Centre, Singapore
  - Tan Tock Seng Hospital, Singapore
- Slovakia (2):
  - Nemocnica s poliklinikou Sv. Jakuba, n.o. Bardejov, Bardejov
  - Univerzitna nemocnica Bratislava, Nemocnica Ruzinov, Bratislava
- South Africa (4):
  - Emery Clinical Services, Alberton, Gauteng
  - University of Pretoria Oncology Department, Pretoria, Gauteng
  - Johese Clinical Research, Pretoria, Gauteng
  - Cape Town Oncology Trials Pty Ltd, Cape Town, Western Cape
- South Korea (19):
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Inje University Haeundae Paik Hospital, Busan, Gyeonggi-do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Kyungpook National University Chilgok Hospital, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (18):
  - Hospital de Mataro, Mataró, Barcelona
  - Hospital Universitario Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Universitario Donostia, Donostia / San Sebastian, Guipuzcoa
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, La Coruña
  - Complejo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Specialist, Barcelona
  - Hospital Universitari Quiron Dexeus, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - ICO Girona - Hospital Universitari de Girona Dr. Josep Trueta, Girona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - MD Anderson Cancer Centre, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Quiron Sagrado Corazon, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Txagorritxu, Vitoria-Gasteiz
- Taiwan (7):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
- Thailand (7):
  - King Chulalongkorn Memorial Hospital, Patumwan, Bangkok
  - Rajavithi Hospital, Rajathevee, Bangkok
  - Srinagarind Hospital, Muang, Changwat Khon Kaen
  - Naresuan University Hospital, Muang, Changwat Phitsanulok
  - Songklanagarind Hospital, Hat Yai, Changwat Songkhla
  - Maharaj Nakorn Chiang Mai Hospital, Muang, Chiang Mai
  - Siriraj Hospital, Bangkok
- Turkey (Türkiye) (19):
  - Acibadem Adana Hospital, Adana
  - Baskent University Adana Application and Research Center, Adana
  - Adana Numune Training and Research Hospital, Adana
  - Cukurova University Medical Faculty, Adana
  - Adana City Hospital, Adana
  - Ankara University Medical Faculty, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Memorial Antalya Hastanesi, Antalya
  - Okmeydani Research and Training Hospital, Istanbul
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Bakirkoy Dr. Sadi Konuk Teaching and Research Hospital, Istanbul
  - Medipol University Medical Faculty, Istanbul
  - Kartal Lutfi Kirdar Research and Training Hospital, Istanbul
  - Ege University Medical Faculty, Izmir
  - Inonu Uni. Med. Fac., Malatya
  - Mersin University Medical Faculty, Mersin
  - Sakarya Traning and Research Hospital, Sakarya
  - Namik Kemal University, Tekirdağ
- Ukraine (16):
  - CI Chernivtsi RC Oncological Dispensary Bukovinian SMU Ch of Oncology and Radiology, Chernivtsi
  - CI Dnipropetrovsk CMCH #4 of Dnipropetrovsk RC Dept of Chemotherapy SI Dnipropetrovsk MA of MOHU, Dnipro
  - CI Transcarpathian Cl Onc Center Dep of Surgery#1 SHEI Ivano-Frankivsk NMU, Ivano-Frankivsk
  - SI S.P.Grygoriev Institute of Medical Radiology of NAMSU, Kharkiv
  - Communal Non-profit Enterprise Regional Center of Oncology, Kharkiv
  - Kherson Regional Oncologic Dispensary, Kherson
  - Treatment-Diagnostic Center of Private Enterprise of PPC Atsynus, Kropyvnytskyi
  - CI Kryvyi Rih Oncological Dispensary of DRC, Kryvyi Rih, Dnipropetrovsk Region
  - Kyiv City Clinical Oncological Center, Kyiv
  - Treatment-Prevention Institution Volyn Regional Oncological Dispensary, Lutsk
  - Lviv State Oncological Regional Treatment and Diagnostic Center, Lviv
  - Odesa Regional Oncologic Dispensary, Odesa
  - RCI Sumy Regional Clinical Oncological Dispensary, Sumy
  - CCCH City Oncological Center SHEI Uzhgorod NU, Uzhhorod
  - Podilskyi Regional Oncological Center, Vinnytsia
  - Vinnytsia Regional Clinical Oncological Dispensary, Vinnytsia
- United Kingdom (6):
  - Southend University Hospital, Westcliff-on-Sea, Essex
  - Cheltenham General Hospital, Cheltenham, Gloucestershire
  - Chelsea and Westminster Hospital, London, Greater London
  - Mount Vernon Hospital, Stevenage, Hertfordshire
  - The Clatterbridge Cancer Centre, Metropolitan Borough of Wirral, Merseyside
  - Royal Stoke University Hospital, Stoke-on-Trent, Staffordshire

REFERENCES:
- [Result] Reck M, Barlesi F, Yang JC, Westeel V, Felip E, Ozguroglu M, Dols MC, Sullivan R, Kowalski DM, Andric Z, Lee DH, Sezer A, Hu P, Wang X, von Heydebreck A, Jacob N, Mehr KT, Park K. Avelumab Versus Platinum-Based Doublet Chemotherapy as First-Line Treatment for Patients With High-Expression Programmed Death-Ligand 1-Positive Metastatic NSCLC: Primary Analysis From the Phase 3 JAVELIN Lung 100 Trial. J Thorac Oncol. 2024 Feb;19(2):297-313. doi: 10.1016/j.jtho.2023.09.1445. Epub 2023 Sep 24. PMID 37748693
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=EMR%20100070-005
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Avelumab Biweekly: Participants received Avelumab at a dose of 10 milligrams per kilogram (mg/kg) as a 1-hour (-10/+20 minutes) intravenous (IV) infusion once every 2 weeks until disease progression or unacceptable toxicities.
- Avelumab Weekly: Participants received Avelumab at a dose of 10 mg/kg as a 1-hour (-10/+20 minutes) IV infusion every week for 12 consecutive weeks, followed by Avelumab at a dose of 10 mg/kg once every 2 weeks until disease progression or unacceptable toxicities.
- Chemotherapy: Participants with tumor of nonsquamous histology received Pemetrexed (500 milligrams per square meter [mg/m^2]) in combination with Cisplatin (75 mg/m^2) administered on Day 1 of each cycle or pemetrexed (500 mg/m^2) in combination with carboplatin (area under the concentration curve [AUC] 6 milligrams per milliliter [mg/mL] * minutes [min] administered on Day 1 of each cycle). Participants who were assigned pemetrexed could continue to receive pemetrexed as a maintenance therapy after 4 cycles of platinum-based chemotherapy if their disease had not progressed, or in accordance with pemetrexed local label. Participants with tumor of squamous histology received Paclitaxel (200 mg/m^2) plus carboplatin (AUC 6 mg/mL * min administered on Day 1 of each cycle) or Gemcitabine (1250 mg/m^2 administered on Day 1 and Day 8 of each cycle) plus cisplatin (75 mg/m^2) or Gemcitabine (1000 mg/m^2 administered on Day 1 and Day 8 of each cycle) plus carboplatin (AUC 5 mg/mL * min) in 3-week cycles up to a maximum of 6 cycles of IV injection or until disease progression or unacceptable toxicities.
Period: Overall Study
Arm/Group | Avelumab Biweekly | Avelumab Weekly | Chemotherapy
Started | 366 | 322 | 526
Completed | 366 | 322 | 526
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Avelumab Biweekly | Avelumab Weekly | Chemotherapy | Total
Number analyzed (Participants) | 366 | 322 | 526 | 1214
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 190 | 168 | 289 | 647
  >=65 years | 176 | 154 | 237 | 567
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 69 | 145 | 298
  Male | 282 | 253 | 381 | 916
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 20 | 38 | 72
  Not Hispanic or Latino | 338 | 296 | 466 | 1100
  Unknown or Not Reported | 14 | 6 | 22 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 85 | 53 | 104 | 242
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 1 | 2 | 4 | 7
  White | 254 | 250 | 375 | 879
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 25 | 17 | 43 | 85

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Assessed by Independent Review Committee (IRC) in High Programmed Death Ligand 1 (PD-L1) + Full Analysis Set (FAS)
Description: PFS is defined as the time from date of randomization until date of the first documentation of progressive disease (PD) or death due to any cause in the absence of documented PD, whichever occurs first. PD is defined as at least a 20 percent (%) increase in the sum of the longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. PFS was measured using Kaplan-Meier (KM) estimates.
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: High PD-L1+ FAS included all high expression PD-L1+ participants who were randomized to study intervention. High expression PD-L1+ participants with greater than or equal to (>=) 80 percent (%) of tumor cells deemed positive for PD-L1 expression at any staining intensity (1+, 2+, or 3+).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab Biweekly | Chemotherapy
Number analyzed (Participants) | 151 | 216
months | 8.4 [5.4 to 12.6] | 5.6 [5.4 to 6.8]
Statistical Analysis 1: Comparison: Avelumab Biweekly vs Chemotherapy; Test type: Superiority; p = 0.0070, Log Rank; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.54 to 0.93]

2. Primary Outcome: Progression Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Assessed by Independent Review Committee (IRC) in High Programmed Death Ligand 1 (PD-L1) + Modified Full Analysis Set (mFAS)
Description: as for outcome 1
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: High PD-L1+ mFAS included all high expression PD-L1+ participants who were randomized to study intervention after weekly Avelumab was included into the randomization allocation. The PDL1+ participants with >= 80% of tumor cells deemed positive for PD-L1 expression at any staining intensity (1+, 2+, or 3+).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab Weekly | Chemotherapy
Number analyzed (Participants) | 130 | 129
months | 7.5 [4.2 to 11.1] | 5.6 [5.0 to 6.8]
Statistical Analysis 1: Comparison: Avelumab Weekly vs Chemotherapy; Test type: Superiority; p = 0.0196, Log Rank; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.52 to 0.98]

3. Primary Outcome: Overall Survival (OS) in High Programmed Death Ligand 1 (PD-L1) + Full Analysis Set (FAS)
Description: OS is defined as the time from randomization to the date of death, regardless of the actual cause of the participant's death. The participants who were still alive at the time of data analysis or who were lost to follow-up OS time was censored at the last recorded date that the participant was known to be alive before the data cutoff date. OS was measured using Kaplan-Meier (KM) estimates.
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab Biweekly | Chemotherapy
Number analyzed (Participants) | 151 | 216
months | 20.1 [15.0 to 24.3] | 14.9 [11.8 to 18.6]
Statistical Analysis 1: Comparison: Avelumab Biweekly vs Chemotherapy; Test type: Superiority; p = 0.1032, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.67 to 1.09]

4. Primary Outcome: Overall Survival (OS) in High Programmed Death Ligand 1 (PD-L1)+ Modified Full Analysis Set (mFAS)
Description: as for outcome 3
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab Weekly | Chemotherapy
Number analyzed (Participants) | 130 | 129
months | 19.3 [14.0 to 28.1] | 15.3 [11.6 to 19.1]
Statistical Analysis 1: Comparison: Avelumab Weekly vs Chemotherapy; Test type: Superiority; p = 0.0630, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.59 to 1.07]

5. Secondary Outcome: Progression Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Assessed by Independent Review Committee (IRC) in Moderate and High Programmed Death Ligand 1 (PD-L1)+ Full Analysis Set (FAS)
Description: as for outcome 1
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: Moderate and High PD-L1+ FAS included all high expression PDL-L1+ participants who were randomized to study intervention. The PD-L1+ participants with >= 50% of tumor cells deemed positive for PD-L1 expression at any staining intensity (1+, 2+, or 3+).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab Biweekly | Chemotherapy
Number analyzed (Participants) | 218 | 304
months | 6.9 [5.4 to 9.6] | 5.6 [5.5 to 6.6]
Statistical Analysis 1: Comparison: Avelumab Biweekly vs Chemotherapy; Test type: Superiority; p = 0.0147, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.62 to 0.98]

6. Secondary Outcome: Progression Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Assessed by Independent Review Committee (IRC) in Moderate and High Programmed Death Ligand 1 (PD-L1)+ Modified Full Analysis Set (mFAS)
Description: as for outcome 1
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: Moderate and High PD-L1+ mFAS included all high expression PD-L1+ participants who were randomized to study intervention after weekly avelumab was included into the randomization allocation. The PD-L1+ participants with >= 50% of tumor cells deemed positive for PD-L1 expression at any staining intensity (1+, 2+, or 3+).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab Weekly | Chemotherapy
Number analyzed (Participants) | 183 | 183
months | 5.6 [2.8 to 8.2] | 5.6 [5.5 to 6.6]
Statistical Analysis 1: Comparison: Avelumab Weekly vs Chemotherapy; Test type: Superiority; p = 0.1753, Log Rank; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.67 to 1.15]

7. Secondary Outcome: Overall Survival (OS) in Moderate and High Programmed Death Ligand 1 (PD-L1)+ Full Analysis Set (FAS)
Description: as for outcome 3
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: Moderate and High PD-L1+ FAS included all high expression PD-L1+ participants who were randomized to study intervention. The PD-L1+ participants with >= 50% of tumor cells deemed positive for PD-L1 expression at any staining intensity (1+, 2+, or 3+).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab Biweekly | Chemotherapy
Number analyzed (Participants) | 218 | 304
months | 18.7 [14.6 to 21.7] | 13.3 [11.4 to 16.6]
Statistical Analysis 1: Comparison: Avelumab Biweekly vs Chemotherapy; Test type: Superiority; p = 0.0257, Log Rank; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.66 to 1.00]

8. Secondary Outcome: Overall Survival (OS) in Moderate and High Programmed Death Ligand 1 (PD-L1)+ Modified Full Analysis Set (mFAS)
Description: as for outcome 3
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab Weekly | Chemotherapy
Number analyzed (Participants) | 183 | 183
months | 16.8 [12.5 to 21.3] | 13.0 [11.1 to 17.0]
Statistical Analysis 1: Comparison: Avelumab Weekly vs Chemotherapy; Test type: Superiority; p = 0.0809, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.66 to 1.07]

9. Secondary Outcome: Overall Survival (OS) in Full Analysis Set (FAS)
Description: as for outcome 3
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: FAS included all participants who were randomized to study intervention.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab Biweekly | Chemotherapy
Number analyzed (Participants) | 366 | 526
months | 15.0 [12.5 to 19.1] | 14.3 [11.8 to 15.6]
Statistical Analysis 1: Comparison: Avelumab Biweekly vs Chemotherapy; Test type: Superiority; p = 0.1294, Log Rank; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.78 to 1.07]

10. Secondary Outcome: Overall Survival (OS) in Modified Full Analysis Set (mFAS)
Description: as for outcome 3
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: mFAS included all participants who were randomized to study intervention after weekly avelumab was included into the randomization allocation.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab Weekly | Chemotherapy
Number analyzed (Participants) | 322 | 321
months | 15.4 [12.1 to 18.1] | 14.8 [11.6 to 16.4]
Statistical Analysis 1: Comparison: Avelumab Weekly vs Chemotherapy; Test type: Superiority; p = 0.2618, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.79 to 1.13]

11. Secondary Outcome: Percentage of Participants With Confirmed Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Independent Review Committee (IRC) in High PD-L1+ Full Analysis Set
Description: Confirmed objective response was defined as the percentage of participants with a confirmed objective response of complete response (CR) or partial response (PR). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions.
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avelumab Biweekly | Chemotherapy
Number analyzed (Participants) | 151 | 216
percentage of participants | 37.7 [30.0 to 46.0] | 30.1 [24.1 to 36.7]
Statistical Analysis 1: Comparison: Avelumab Biweekly vs Chemotherapy; Test type: Superiority; p = 0.0640, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.91 to 2.18]

12. Secondary Outcome: Percentage of Participants With Confirmed Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Independent Review Committee (IRC) in High PD-L1+ Modified Full Analysis Set
Description: as for outcome 11
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avelumab Weekly | Chemotherapy
Number analyzed (Participants) | 130 | 129
percentage of participants | 34.6 [26.5 to 43.5] | 30.2 [22.5 to 38.9]
Statistical Analysis 1: Comparison: Avelumab Weekly vs Chemotherapy; Test type: Superiority; p = 0.2217, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.73 to 2.07]

13. Secondary Outcome: Percentage of Participants With Confirmed Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Independent Review Committee (IRC) in Moderate and High PD-L1+ Full Analysis Set
Description: as for outcome 11
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avelumab Biweekly | Chemotherapy
Number analyzed (Participants) | 218 | 304
percentage of participants | 33.5 [27.3 to 40.2] | 30.3 [25.1 to 35.8]
Statistical Analysis 1: Comparison: Avelumab Biweekly vs Chemotherapy; Test type: Superiority; p = 0.1912, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.81 to 1.72]

14. Secondary Outcome: Percentage of Participants With Confirmed Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Independent Review Committee (IRC) in Moderate and High PD-L1+ Modified Full Analysis Set
Description: as for outcome 11
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avelumab Weekly | Chemotherapy
Number analyzed (Participants) | 183 | 183
percentage of participants | 30.6 [24.0 to 37.8] | 30.6 [24.0 to 37.8]
Statistical Analysis 1: Comparison: Avelumab Weekly vs Chemotherapy; Test type: Superiority; p = 0.4951, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.64 to 1.57]

15. Secondary Outcome: Duration of Response (DOR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Independent Review Committee (IRC) in High Programmed Death Ligand 1 (PD-L1)+ Full Analysis Set (FAS)
Description: DOR was defined for participants with confirmed response, as the time from first documentation of objective response (Complete Response [CR] or Partial Response [PR]) to the date of first documentation of progression disease (PD) or death due to any cause, whichever occurred first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the SLD of all lesions. PD: At least a 20 percent (%) increase in the sum of the longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: High PD-L1+ FAS was used. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Avelumab Biweekly | Chemotherapy
Number analyzed (Participants) | 57 | 65
months | 35.9 [1.4 to 60.8] | 8.4 [1.0 to 63.9]

16. Secondary Outcome: Duration of Response (DOR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Independent Review Committee (IRC) in High Programmed Death Ligand 1 (PD-L1)+ Modified Full Analysis Set (mFAS)
Description: as for outcome 15
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: High PD-L1+ mFAS was used. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Avelumab Weekly | Chemotherapy
Number analyzed (Participants) | 45 | 39
months | 19.4 [3.8 to 43.9] | 8.4 [1.0 to 35.9]

17. Secondary Outcome: Change From Baseline in European Quality Of Life 5-dimensions (EQ-5D-5L) Visual Analog Scale (VAS) in High PD-L1+ Health-related Quality of Life (HRQoL) Analysis Set at End of Treatment
Description: EQ-5D-5L is comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive overall score using a visual analog scale (VAS) that ranged from 0 to 100 millimeter (mm), where 0 is the worst health you can imagine and 100 is the best health you can imagine.
Time Frame: Baseline, End of treatment (up to Week 283.9)
Population: High PD-L1+HRQoL analysis set includes all high expression PD-L1+ FAS participants who have 1 baseline HRQoL assessment and have >=1 post-baseline HRQoL questionnaire complete. The high expression PDL1+ participants were with >= 80% of tumor cells deemed positive for PD-L1 expression at any staining intensity (1+, 2+, or 3+). Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Avelumab Biweekly | Chemotherapy
Number analyzed (Participants) | 56 | 107
millimeter (mm) | -6.2 (23.61) | -5.2 (20.48)

18. Secondary Outcome: Change From Baseline in European Quality Of Life 5-dimensions (EQ-5D-5L) Visual Analog Scale (VAS) in High Programmed Death Ligand 1 (PD-L1)+ Modified HRQoL Analysis Set
Description: as for outcome 17
Time Frame: Baseline, End of treatment (Week 283.9)
Population: High PD-L1+ Modified HRQoL Analysis Set included all mFAS participants who have 1 baseline HRQoL assessment and have >=1 post-baseline HRQoL questionnaire completed. The high expression PDL1+ participants were with >= 80% of tumor cells deemed positive for PD-L1 expression at any staining intensity (1+, 2+, or 3+). Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Avelumab Weekly | Chemotherapy
Number analyzed (Participants) | 53 | 70
millimeter | -10.3 (22.49) | -3.9 (20.21)

19. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life (EORTC QLQ-C30) Global Health Status at End of Treatment (EOT) in High Programmed Death Ligand 1 (PD-L1)+ HRQoL Analysis Set
Description: EORTC QLQ-C30 was a 30-question tool used to assess the overall quality of life (QoL) in cancer participants. It consisted of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, role, cognitive, emotional, social), and 9 symptom scales/items (Fatigue, nausea and vomiting, pain, dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, financial impact). The EORTC QLQ-C30 GHS/QoL score ranged from 0 to 100; High score indicated better GHS/QoL. Score 0 represents: very poor physical condition and QoL. Score 100 represents: excellent overall physical condition and QoL.
Time Frame: Baseline, End of treatment (up to Week 283.9)
Population: High PD-L1+HRQoL analysis set includes all high expression PD-L1 FAS participants who have 1 baseline HRQoL assessment and have >=1 post-baseline HRQoL questionnaire complete. The high expression PDL1+ participants were with >= 80% of tumor cells deemed positive for PD-L1 expression at any staining intensity (1+, 2+, or 3+).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Avelumab Biweekly | Chemotherapy
Number analyzed (Participants) | 56 | 108
score on a scale | -0.3 (22.30) | -6.1 (24.55)

20. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life (EORTC QLQ-C30) Global Health Status at End of Treatment (EOT) in High Programmed Death Ligand 1 (PD-L1)+ Modified HRQoL Analysis Set
Description: as for outcome 19
Time Frame: Baseline, End of treatment (Week 283.9)
Population: High PD-L1+modified HRQoL analysis set includes all high expression PD-l1+ mFAS participants who have 1 baseline HRQoL assessment and have ≥1 post-baseline HRQoL questionnaire completed. The high expression PDL1+ participants were with >= 80% of tumor cells deemed positive for PD-L1 expression at any staining intensity (1+, 2+, or 3+). Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Avelumab Weekly | Chemotherapy
Number analyzed (Participants) | 53 | 71
score on a scale | -12.9 (21.03) | -4.5 (23.30)

21. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer 13 (EORTC QLQ-LC13) at End of Treatment (EOT) in High Programmed Death Ligand 1 (PD-L1)+ HRQoL Analysis Set
Description: EORTC QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy. The EORTC QLQ-LC13 module generated one multiple-item score assessing dyspnea and a series of single item scores assessing coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, pain in chest, pain in arms or shoulder and pain in other parts. Score range: 0 (no burden of symptom domain or single symptom item) to 100 (highest burden of symptoms for symptom domains and single items).
Time Frame: Baseline, End of treatment (up to Week 283.9)
Population: High PD-L1+ HRQoL analysis set includes all high expression PD-L1+ FAS participants who have 1 baseline HRQoL assessment and have >=1 post-baseline HRQoL questionnaire complete. The high expression PDL1+ participants were with >= 80% of tumor cells deemed positive for PD-L1 expression at any staining intensity (1+, 2+, or 3+). Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Avelumab Biweekly | Chemotherapy
Number analyzed (Participants) | 56 | 108
score on a scale
  Dyspnea | 7.3 (24.10) | 5.2 (19.66)
  Coughing | 2.4 (29.04) | -4.3 (27.01)
  Hemoptysis | -1.8 (21.48) | 1.5 (13.95)
  Sore mouth | 3.0 (18.28) | 1.9 (21.77)
  Dysphagia | 3.0 (19.36) | -0.6 (21.36)
  Peripheral neuropathy | 3.6 (17.60) | 10.8 (24.46)
  Alopecia | 0.0 (8.98) | 14.2 (32.93)
  Pain in chest | -4.2 (22.96) | -1.5 (26.33)
  Pain in arm or shoulder | 0.6 (32.71) | 1.9 (26.50)
  Pain in other parts | 1.8 (33.29) | 1.5 (30.36)

22. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer 13 (EORTC QLQ-LC13) at End of Treatment (EOT) in High Programmed Death Ligand 1 (PD-L1)+ Modified HRQoL Analysis Set
Description: as for outcome 21
Time Frame: Baseline, End of treatment (up to Week 283.9)
Population: High PD-L1+ modified HRQoL analysis set was used. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Avelumab Weekly | Chemotherapy
Number analyzed (Participants) | 53 | 71
score on a scale
  Dyspnea | 6.1 (27.19) | 4.9 (18.77)
  Coughing | -0.6 (28.87) | -5.2 (24.34)
  Hemoptysis | -0.6 (17.89) | 0.0 (12.59)
  Sore mouth: number analyzed (Participants) | 52 | 71
  Sore mouth | 0.6 (13.97) | 1.9 (17.71)
  Dysphagia | 3.8 (14.10) | -0.5 (22.88)
  Peripheral neuropathy | 0.6 (21.17) | 9.9 (23.49)
  Alopecia | -2.5 (17.11) | 15.0 (29.70)
  Pain in chest | 2.5 (29.13) | -0.5 (25.50)
  Pain in arm or shoulder | 4.4 (30.69) | 1.4 (25.46)
  Pain in other parts | 10.1 (28.93) | 1.4 (28.97)

23. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and AEs of Special Interest (AESIs)
Description: Adverse event (AE) was defined as any untoward medical occurrence in a participant, which does not necessarily have causal relationship with treatment. A serious AE was defined as an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged in participant hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. The term TEAEs were those events with onset dates occurring during the on-treatment period or if the worsening of an event is during the on-treatment period TEAEs included both serious TEAEs and non-serious TEAEs. Any AE that was suspicious to be a potential Immune-related adverse event (irAE) including infusion related reactions were considered AESIs. Number of participants with TEAEs and AESIs were reported.
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: The Safety analysis set (Safety-AS) included all randomized participants who were administered at least one dose of the study medication, that is (i.e.) avelumab or chemotherapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab Biweekly | Avelumab Weekly | Chemotherapy
Number analyzed (Participants) | 361 | 318 | 500
Participants
  TEAEs | 346 | 308 | 484
  AESIs | 158 | 160 | 173

24. Secondary Outcome: Number of Participants With Shift From Baseline to Greater Than or Equal to (>=) Grade 3 in Laboratory Parameter Values Based on National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.03
Description: Number of participants with shifts from Baseline values (Grade 0/1/2/3) to abnormal post-baseline values (shift to >= Grade 4) were reported as per NCI-CTCAE, v4.03 graded from Grade 1 to 5. Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening; Grade 5: Death. Shifts in laboratory parameter (anemia, lymphocyte count decreased, neutrophil count decreased, platelet count decreased, white blood cell count decreased, alanine aminotransferase increased, alkaline phosphatase increased, aspartate aminotransferase increased, blood bilirubin increased, creatine phosphokinase increased, creatinine increased and Hyperglycemia) were reported.
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab Biweekly | Avelumab Weekly | Chemotherapy
Number analyzed (Participants) | 361 | 318 | 500
Participants
  Anemia: Grade 0 to Grade 3 | 4 | 2 | 58
  Anemia: Grade 1 to Grade 3 | 4 | 5 | 30
  Anemia: Grade 2 to Grade 3 | 4 | 6 | 6
  Lymphocyte count decreased: Grade 0 to Grade 3 | 16 | 15 | 31
  Lymphocyte count decreased: Grade 0 to Grade 4 | 1 | 2 | 3
  Lymphocyte count decreased: Grade 1 to Grade 3 | 2 | 10 | 12
  Lymphocyte count decreased: Grade 2 to Grade 3 | 7 | 6 | 12
  Lymphocyte count decreased: Grade 2 to Grade 4 | 0 | 0 | 1
  Lymphocyte count decreased: Grade 3 to Grade 4 | 0 | 0 | 1
  Neutrophil count decreased: Grade 0 to Grade 3 | 4 | 4 | 65
  Neutrophil count decreased: Grade 0 to Grade 4 | 0 | 3 | 25
  Neutrophil count decreased: Grade 1 to Grade 3 | 1 | 0 | 1
  Platelet count decreased: Grade 0 to Grade 3 | 0 | 1 | 18
  Platelet count decreased: Grade 0 to Grade 4 | 0 | 3 | 20
  Platelet count decreased: Grade 1 to Grade 3 | 0 | 1 | 0
  White blood cell count decreased: Grade 0 to Grade 3 | 0 | 3 | 24
  White blood cell count decreased: Grade 0 to Grade 4 | 0 | 1 | 11
  Alanine aminotransferase increased: Grade 0 to Grade 3 | 12 | 8 | 5
  Alanine aminotransferase increased: Grade 0 to Grade 4 | 1 | 1 | 3
  Alanine aminotransferase increased: Grade 1 to Grade 3 | 1 | 0 | 2
  Alkaline phosphatase increased: Grade 0 to Grade 3 | 0 | 3 | 1
  Alkaline phosphatase increased: Grade 1 to Grade 3 | 1 | 3 | 1
  Alkaline phosphatase increased: Grade 1 to Grade 4 | 0 | 0 | 1
  Alkaline phosphatase increased: Grade 2 to Grade 3 | 0 | 1 | 0
  Aspartate aminotransferase increased: Grade 0 to Grade 3 | 7 | 4 | 3
  Aspartate aminotransferase increased: Grade 0 to Grade 4 | 1 | 2 | 2
  Aspartate aminotransferase increased: Grade 1 to Grade 3 | 0 | 0 | 1
  Blood bilirubin increased: Grade 0 to Grade 3 | 0 | 4 | 3
  Blood bilirubin increased: Grade 0 to Grade 4 | 0 | 1 | 0
  Creatine phosphokinase increased: Grade 0 to Grade 3 | 6 | 5 | 1
  Creatine phosphokinase increased: Grade 0 to Grade 4 | 5 | 0 | 0
  Creatine phosphokinase increased: Grade 1 to Grade 4 | 0 | 1 | 0
  Creatine phosphokinase increased: Grade 2 to Grade 3 | 0 | 1 | 0
  Creatinine increased: Grade 0 to Grade 3 | 6 | 4 | 4
  Creatinine increased: Grade 1 to Grade 3 | 0 | 0 | 1
  Hyperglycemia: Grade 0 to Grade 3 | 21 | 20 | 35
  Hyperglycemia: Grade 0 to Grade 4 | 0 | 0 | 3

25. Secondary Outcome: Number of Participants With Maximal On-Treatment Changes From Baseline in Vital Signs - Maximal Body Temperature Increase
Description: The number of participants with changes from baseline in increased Body Temperature (degree Celsius [°C]) were reported by using criteria: Baseline temperature (temp.) less than (<) 37°C, on treatment change <1°C, 1 - <2°C, 2 - <3°C, greater than or equal to (>=)3°C and missing; Baseline temp. 37 - <38°C, on treatment change <1°C, 1 - <2°C, 2 - <3°C, >=3°C and missing; Baseline temp. 38 - <39°C, on treatment change <1°C, 1 - <2°C, 2 - <3°C, >=3°C and missing; Baseline temp. 39-<40°C, on treatment change <1°C, 1 - <2°C, 2 - <3°C, >=3°C and missing; Baseline temp. >=40°C, on treatment change <1°C, 1 - <2°C, 2 - <3°C, >=3°C and missing; Baseline temp. missing, on treatment change missing.
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab Biweekly | Avelumab Weekly | Chemotherapy
Number analyzed (Participants) | 361 | 318 | 500
Participants
  Baseline temp. <37°C, on treatment change <1°C | 271 | 256 | 403
  Baseline temp.<37°C, on treatment change 1 - <2°C | 45 | 32 | 33
  Baseline temp. <37°C, on treatment change 2 - <3°C | 3 | 2 | 0
  Baseline temp. <37°C, on treatment change >=3°C | 0 | 1 | 0
  Baseline temp. <37°C, on treatment change missing | 16 | 6 | 21
  Baseline temp. 37 - <38°C, on treatment change <1°C | 23 | 19 | 37
  Baseline temp. 37 - <38°C, on treatment change 1 - <2°C | 1 | 2 | 1
  Baseline temp. 37 - <38°C, on treatment change 2 - <3°C | 0 | 0 | 0
  Baseline temp. 37 - <38°C, on treatment change >=3°C | 0 | 0 | 0
  Baseline temp. 37 - <38°C, on treatment change missing | 1 | 0 | 3
  Baseline temp. 38 - <39°C, on treatment change <1°C | 0 | 0 | 0
  Baseline temp. 38 - <39°C, on treatment change 1 - <2°C | 0 | 0 | 0
  Baseline temp. 38 - <39°C, on treatment change 2 - <3°C | 0 | 0 | 0
  Baseline temp. 38 - <39°C, on treatment change >=3°C | 0 | 0 | 0
  Baseline temp. 38 - <39°C, on treatment change missing | 0 | 0 | 0
  Baseline temp. 39 - <40°C, on treatment change <1°C | 1 | 0 | 0
  Baseline temp. 39 - <40°C, on treatment change 1 - <2°C | 0 | 0 | 0
  Baseline temp. 39 - <40°C, on treatment change 2 - <3°C | 0 | 0 | 0
  Baseline temp. 39 - <40°C, on treatment change >=3°C | 0 | 0 | 0
  Baseline temp. 39 - <40°C, on treatment change missing | 0 | 0 | 0
  Baseline temp. >=40°C, on treatment change <1°C | 0 | 0 | 0
  Baseline temp. >=40°C, on treatment change 1 - <2°C | 0 | 0 | 0
  Baseline temp. >=40°C, on treatment change 2 - <3°C | 0 | 0 | 0
  Baseline temp. >=40°C, on treatment change >=3°C | 0 | 0 | 0
  Baseline temp. >=40°C, on treatment change missing | 0 | 0 | 0
  Baseline temp. missing, on treatment change missing | 0 | 0 | 2

26. Secondary Outcome: Number of Participants With Maximal On-Treatment Changes From Baseline in Vital Signs - Maximal Weight Increase/Decrease
Description: The number of participants with maximal on-treatment changes from baseline in Increase (Ic.)/Decrease (Dc.) in maximal weight were reported by using criteria: Ic./Dc. From baseline, on treatment (TR) change <10 percentage (%), >=10% and missing.
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab Biweekly | Avelumab Weekly | Chemotherapy
Number analyzed (Participants) | 361 | 318 | 500
Participants
  Ic. from baseline, on TR change <10% | 302 | 280 | 436
  Ic. from baseline, on TR change >=10% | 38 | 28 | 39
  Ic. from baseline, on TR change missing | 21 | 10 | 25
  Dc. from baseline, on TR change <10% | 296 | 258 | 423
  Dc. from baseline, on TR change >=10% | 44 | 50 | 52
  Dc. from baseline, on TR change missing | 21 | 10 | 25

27. Secondary Outcome: Number of Participants With Maximal On-Treatment Changes From Baseline in Vital Signs - Maximal Heart Rate Increase/Decrease
Description: The number of participants with maximal on-treatment (TR) changes from baseline (BS) in Increase (Ic.)/Decrease (Dc.) heart rate (HR) (beats per minute [bpm]) were reported by using criteria: Ic./Dc. BS HR <100/>=100 bpm, on treatment change =<20 bpm, >20 - =<40 bpm, >40 bpm and missing; Ic./Dc. BS HR missing, on treatment change missing.
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab Biweekly | Avelumab Weekly | Chemotherapy
Number analyzed (Participants) | 361 | 318 | 500
Participants
  Ic. BS HR <100 bpm, on TR change =<20 bpm | 206 | 202 | 332
  Ic. BS HR <100 bpm, on TR change >20 - =<40 bpm | 86 | 66 | 85
  Ic. BS HR <100 bpm, on TR change >40 bpm | 21 | 12 | 9
  Ic. BS HR <100 bpm, on TR change missing | 14 | 5 | 16
  Ic. BS HR >= 100 bpm, on TR change =<20 bpm | 31 | 30 | 46
  Ic. BS HR >= 100 bpm, on TR change >20 - =<40 bpm | 0 | 2 | 3
  Ic. BS HR >= 100 bpm, on TR change >40 bpm | 0 | 0 | 0
  Ic. BS HR >= 100 bpm, on TR change missing | 3 | 1 | 7
  Ic. BS HR missing, on TR change missing | 0 | 0 | 2
  Dc. BS HR <100 bpm, on TR change =<20 bpm | 267 | 227 | 385
  Dc. BS HR <100 bpm, on TR change >20 - =<40 bpm | 44 | 52 | 40
  Dc. BS HR <100 bpm, on TR change >40 bpm | 2 | 1 | 1
  Dc. BS HR <100 bpm, on TR change missing | 14 | 5 | 16
  Dc. BS HR >= 100 bpm, on TR change =<20 bpm | 14 | 13 | 20
  Dc. BS HR >= 100 bpm, on TR change >20 - =<40 bpm | 6 | 12 | 26
  Dc. BS HR >= 100 bpm, on TR change >40 bpm | 11 | 7 | 3
  Dc. BS HR >= 100 bpm, on TR change missing | 3 | 1 | 7
  Dc. BS HR missing, on TR change missing | 0 | 0 | 2

28. Secondary Outcome: Number of Participants With Maximal On-Treatment Changes From Baseline in Vital Signs - Maximal Systolic Blood Pressure Increase/Decrease and Maximal Diastolic Blood Pressure Increase/Decrease
Description: The number of participants with maximal on-treatment changes from baseline (BS) in Increase (Ic.)/Decrease (Dc.) Systolic Blood Pressure (SBP) and diastolic blood pressure (DBP) (millimeter of mercury [mmHg]) were reported by using criteria: Ic./Dc. BS SBP <140 mmHg and >=140 mmHg, on maximal treatment (TR) change =<20 mmHg, >20 - =<40 mmHg, >40 mmHg and missing; Ic./Dc. BS SBP missing, on maximal treatment (TR) change missing; Ic./Dc. BS DBP <90 mmHg and >= 90 mmHg, on maximal TR change =<20 mmHg, >20 - =<40 mmHg, >40 mmHg and missing; Ic./Dc. BS DBP missing on maximal TR change missing.
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab Biweekly | Avelumab Weekly | Chemotherapy
Number analyzed (Participants) | 361 | 318 | 500
Participants
  Ic. BS SBP <140 mmHg, on TR change =<20 mmHg | 219 | 209 | 278
  Ic. BS SBP <140 mmHg, on TR change >20 - =<40 mmHg | 61 | 56 | 104
  Ic. BS SBP <140 mmHg, on TR change >40 mmHg | 16 | 16 | 10
  Ic. BS SBP <140 mmHg, on TR change missing | 14 | 4 | 21
  Ic. BS SBP >=140 mmHg, on TR change =<20 mmHg | 41 | 26 | 78
  Ic. BS SBP >=140 mmHg, on TR change >20 - =<40 mmHg | 7 | 5 | 5
  Ic. BS SBP >=140 mmHg, on TR change >40 mmHg | 0 | 0 | 1
  Ic. BS SBP > = 140 mmHg, on TR change missing | 3 | 2 | 2
  Ic. BS SBP missing, on TR change missing | 0 | 0 | 1
  Dc. BS SBP <140 mmHg, on TR change =<20 mmHg | 220 | 204 | 322
  Dc. BS SBP <140 mmHg, on TR change >20 - =<40 mmHg | 70 | 70 | 69
  Dc. BS SBP <140 mmHg, on TR change >40 mmHg | 6 | 7 | 1
  Dc. BS SBP <140 mmHg, on TR change missing | 14 | 4 | 21
  Dc. BS SBP >=140 mmHg, on TR change =<20 mmHg | 11 | 6 | 32
  Dc. BS SBP >=140 mmHg, on TR change >20 - =<40 mmHg | 25 | 15 | 34
  Dc. BS SBP >=140 mmHg, on TR change >40 mmHg | 12 | 10 | 18
  Dc. BS SBP > = 140 mmHg, on TR change missing | 3 | 2 | 2
  Dc. BS SBP missing, on TR change missing | 0 | 0 | 1
  Ic. BS DBP <90 mmHg, on TR change =<20 mmHg | 272 | 260 | 402
  Ic. BS DBP <90 mmHg, on TR change >20 - =<40 mmHg | 48 | 37 | 45
  Ic. BS DBP <90 mmHg, on TR change >40 mmHg | 0 | 1 | 1
  Ic. BS DBP <90 mmHg, on TR change missing | 17 | 5 | 23
  Ic. BS DBP missing, on TR change missing | 0 | 0 | 1
  Ic. BS DBP >=90 mmHg, on TR change =<20 mmHg | 24 | 12 | 28
  Ic. BS DBP >=90 mmHg, on TR change >20 - =<40 mmHg | 0 | 1 | 0
  Ic. BS DBP >=90 mmHg, on TR change >40 mmHg | 0 | 1 | 0
  Ic. BS DBP >=90 mmHg, on TR change missing | 0 | 1 | 0
  Dc. BS DBP <90 mmHg, on TR change =<20 mmHg | 279 | 264 | 415
  Dc. BS DBP <90 mmHg, on TR change >20 - =<40 mmHg | 38 | 33 | 32
  Dc. BS DBP <90 mmHg, on TR change >40 mmHg | 3 | 1 | 1
  Dc. BS DBP <90 mmHg, on TR change missing | 17 | 5 | 23
  Dc. BS DBP >=90 mmHg, on TR change =<20 mmHg | 11 | 5 | 18
  Dc. BS DBP >=90 mmHg,on TR change >20 - =<40 mmHg | 12 | 9 | 10
  Dc. BS DBP >=90 mmHg, on TR change >40 mmHg | 1 | 0 | 0
  Dc. BS DBP >=90 mmHg, on TR change missing | 0 | 1 | 0
  Dc. BS DBP missing, on TR change missing | 0 | 0 | 1

29. Secondary Outcome: Number of Participants With Maximal On-Treatment Changes From Baseline in Vital Signs - Maximal Respiration Rate Increase/Decrease
Description: The number of participants with maximal on-treatment (TR) changes from baseline (BS) in Increase (Ic.)/Decrease (Dc.) maximal Respiration Rate (RR) were reported by using criteria: Ic./Dc. BS RR <20 breaths per minute (breaths/min), on TR change =<5 breaths/min, >5 - =<10 breaths/min, >10 breaths/min and missing. Ic./Dc. BS RR missing, on TR change missing. Ic./Dc. BS RR >=20 breaths/min, on TR change =<5 breaths/min, >5 - =<10 breaths/min, >10 breaths/min and missing.
Time Frame: Time from date of randomization up to data cutoff (assessed up to 71.5 months)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab Biweekly | Avelumab Weekly | Chemotherapy
Number analyzed (Participants) | 361 | 318 | 500
Participants
  Ic. BS RR <20 breaths/min, on TR change =<5 breaths/min | 221 | 224 | 306
  Ic.BS RR<20 breaths/min, on TR change >5 - = <10 breaths/min | 18 | 13 | 26
  Ic. BS RR <20 breaths/min, on TR change >10 breaths/min | 1 | 1 | 2
  Ic. BS RR <20 breaths/min, on TR change missing | 11 | 4 | 14
  Ic. BS RR >=20 breaths/min, on TR change =<5 breaths/min | 89 | 68 | 124
  Ic.BS RR >=20 breaths/min, on TR change >5 - =<10 breaths/min | 5 | 4 | 2
  Ic. BS RR >=20 breaths/min, on TR change >10 breaths/min | 3 | 1 | 0
  Ic. BS RR >=20 breaths/min, on TR change missing | 7 | 2 | 15
  Ic. BS RR missing, on TR change missing | 6 | 1 | 11
  Dc. BS RR <20 breaths/min, on TR change =<5 breaths/min | 232 | 236 | 325
  Dc. BS RR <20 breaths/min, on TR change >5 - =<10 breaths/min | 8 | 2 | 8
  Dc. BS RR <20 breaths/min, on TR change >10 breaths/min | 0 | 0 | 1
  Dc. BS RR <20 breaths/min, on TR change missing | 11 | 4 | 14
  Dc. BS RR >=20 breaths/min, on TR ch =<5 breaths/min | 79 | 58 | 101
  Dc.BS RR >=20 breaths/min, on TR change >5 - =<10 breaths/min | 14 | 13 | 22
  Dc. BS RR >=20 breaths/min, on TR change >10 breaths/min | 4 | 2 | 3
  Dc. BS RR >=20 breaths/min, on TR change missing | 7 | 2 | 15
  Dc. BS RR missing, on TR change missing | 6 | 1 | 11

30. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities (PCSA) in Electrocardiogram (ECG) Parameters
Description: ECG parameters included heart rate, PR interval, QRS interval, corrected QT interval using Bazett's formula (QTcB) and corrected QT interval using Fridericia's formula (QTcF). PCSA criteria for abnormal value of ECG parameters: any heart rate <= 50 bpm and decrease from baseline >=20 bpm , any hear rate >= 120 bpm and increase from baseline >= 20 bpm; PR interval: >= 220 milliseconds (ms) and increase from baseline >= 20 ms; QRS interval >= 120 ms; QTcF > 450 ms, > 480 ms, > 500 ms, QTcF increase from baseline > 30 ms and QTcF increase from baseline > 60 ms; QTcB > 450 ms, > 480 ms, > 500 ms, QTcB increase from baseline > 30 ms and QTcB increase from baseline > 60 ms.
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: The Safety analysis set (Safety-AS) included all randomized participants who were administered at least one dose of the study medication, that is (i.e.) avelumab or chemotherapy. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab Biweekly | Avelumab Weekly | Chemotherapy
Number analyzed (Participants) | 264 | 223 | 399
Participants
  Heart Rate <= 50 bpm and decrease from baseline >= 20 bpm | 1 | 1 | 0
  Heart Rate >= 120 bpm and decrease from baseline >= 20 bpm | 10 | 6 | 7
  PR interval >= 220 ms and increase from baseline >= 20 ms | 0 | 5 | 3
  QRS interval >= 120 ms | 18 | 10 | 15
  QTcF > 450 ms | 19 | 13 | 24
  QTcF > 480 ms | 5 | 4 | 11
  QTcF > 500 ms | 3 | 1 | 5
  QTcF increase from baseline > 30 ms | 20 | 12 | 39
  QTcF increase from baseline > 60 ms | 6 | 1 | 13
  QTcB > 450 ms | 49 | 31 | 70
  QTcB > 480 ms | 13 | 11 | 24
  QTcB > 500 ms | 6 | 5 | 16
  QTcB increase from baseline > 30 ms | 32 | 25 | 49
  QTcB increase from baseline > 60 ms | 11 | 7 | 19

31. Secondary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance: Baseline Score Versus (Vs) Worst Post-baseline Score
Description: ECOG performance status measured to assess participant's performance status on a scale of 0 to 5, where 0 = Fully active, able to carry on all pre-disease activities without restriction; 1 = Restricted in physically strenuous activity, ambulatory and able to carry out light or sedentary work; 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; 3 = Capable of only limited self-care, confined to bed/chair for more than 50 percent of waking hours; 4 = Completely disabled, cannot carry on any self-care, totally confined to bed/chair; 5 = dead. ECOG performance status was reported in terms of number of participants with baseline value vs worst post-baseline value (that is [i.e.] highest score).
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab Biweekly | Avelumab Weekly | Chemotherapy
Number analyzed (Participants) | 361 | 318 | 500
Participants
  Baseline score 0, worst post-baseline score 0 | 50 | 35 | 84
  Baseline score 0, worst post-baseline score 1 | 56 | 49 | 83
  Baseline score 0, worst post-baseline score 2 | 8 | 9 | 11
  Baseline score 0, worst post-baseline score 3 | 1 | 7 | 4
  Baseline score 0, worst post-baseline score 4 | 1 | 0 | 0
  Baseline score 0, worst post-baseline score 5 | 0 | 0 | 1
  Baseline score 0, worst post-baseline score Missing | 6 | 4 | 4
  Baseline score 1, worst post-baseline score 0 | 1 | 2 | 4
  Baseline score 1, worst post-baseline score 1 | 168 | 153 | 233
  Baseline score 1, worst post-baseline score 2 | 35 | 32 | 46
  Baseline score 1, worst post-baseline score 3 | 16 | 18 | 6
  Baseline score 1, worst post-baseline score 4 | 3 | 1 | 4
  Baseline score 1, worst post-baseline score 5 | 5 | 1 | 3
  Baseline score 1, worst post-baseline score Missing | 10 | 6 | 16
  Baseline score >=2, worst post-baseline score 0 | 0 | 0 | 0
  Baseline score >=2, worst post-baseline score 1 | 0 | 0 | 0
  Baseline score >=2, worst post-baseline score 2 | 0 | 0 | 0
  Baseline score >=2, worst post-baseline score 3 | 1 | 0 | 0
  Baseline score >=2, worst post-baseline score 4 | 0 | 0 | 0
  Baseline score >=2, worst post-baseline score 5 | 0 | 1 | 0
  Baseline score >=2, worst post-baseline score missing | 0 | 0 | 0
  Baseline score missing, worst post-baseline score 0 | 0 | 0 | 0
  Baseline score missing, worst post-baseline score 1 | 0 | 0 | 1
  Baseline score missing, worst post-baseline score 2 | 0 | 0 | 0
  Baseline score missing, worst post-baseline score 3 | 0 | 0 | 0
  Baseline score missing, worst post-baseline score 4 | 0 | 0 | 0
  Baseline score missing, worst post-baseline score 5 | 0 | 0 | 0
  Baseline score missing, worst post-baseline score missing | 0 | 0 | 0

32. Secondary Outcome: Number of Participants With At Least One Positive Anti-Drug Antibodies (ADAs) and Neutralizing Antibodies (NAbs) for Avelumab
Description: Serum samples were analyzed by a validated electrochemiluminesce immunoassay to detect the presence of antidrug antibodies (ADA). Samples that screened positive were subsequently tested in a confirmatory assay were tested for neutralizing antibodies (nAb). Number of participants with ADA or nAb positive results for Avelumab were reported.
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Population: The Safety analysis set (Safety-AS) included all randomized participants who were administered at least one dose of the study medication, that is (i.e.) avelumab. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab Biweekly | Avelumab Weekly
Number analyzed (Participants) | 360 | 318
Participants
  ADAs to Avelumab | 66 | 38
  NAbs to Avelumab | 43 | 18

ADVERSE EVENTS:
Time Frame: Time from date of randomization up to data cutoff (assessed up to approximately 71.5 months)
Description: Only participants who received study medication were included in the analysis of adverse events. All randomized participants were included in the analysis of all-cause mortality.
Arm/Group | Avelumab Biweekly | Avelumab Weekly | Chemotherapy
All-Cause Mortality (participants affected / at risk) | 279/366 | 237/322 | 405/526
Serious Adverse Events (participants affected / at risk) | 181/361 | 143/318 | 195/500
Other Adverse Events (participants affected / at risk) | 331/361 | 298/318 | 474/500
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab Biweekly (N=361) | Avelumab Weekly (N=318) | Chemotherapy (N=500)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 | 3 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 | 5 | 8
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 6
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 3
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 2
Pneumonia (Infections and infestations) | 28 | 13 | 28
Respiratory tract infection (Infections and infestations) | 4 | 1 | 3
Sepsis (Infections and infestations) | 4 | 1 | 4
Bronchitis (Infections and infestations) | 2 | 5 | 1
Septic shock (Infections and infestations) | 0 | 0 | 6
Disease progression (General disorders) | 33 | 18 | 22
Fatigue (General disorders) | 4 | 0 | 1
Asthenia (General disorders) | 2 | 1 | 5
Pyrexia (General disorders) | 1 | 3 | 8
Infusion related reaction (Injury, poisoning and procedural complications) | 11 | 7 | 0
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 3
Vomiting (Gastrointestinal disorders) | 2 | 0 | 9
Cerebral infarction (Nervous system disorders) | 4 | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 6 | 2
Platelet count decreased (Investigations) | 0 | 0 | 7
Anaemia (Blood and lymphatic system disorders) | 4 | 2 | 19
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 13
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 6
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 5
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 0 | 2
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 | 0 | 0
Amoebiasis (Infections and infestations) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 2 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 0
Influenza (Infections and infestations) | 1 | 2 | 2
Lung abscess (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 3
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Enterobacter infection (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1
Large intestine infection (Infections and infestations) | 0 | 0 | 1
Nosocomial infection (Infections and infestations) | 0 | 0 | 1
Oral fungal infection (Infections and infestations) | 0 | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 2
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0
Sepsis syndrome (Infections and infestations) | 0 | 0 | 1
Systemic candida (Infections and infestations) | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Death (General disorders) | 2 | 2 | 2
Chest pain (General disorders) | 1 | 0 | 1
Sudden death (General disorders) | 1 | 3 | 1
General physical health deterioration (General disorders) | 0 | 3 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 2
Peripheral swelling (General disorders) | 0 | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 1 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 2
Colitis (Gastrointestinal disorders) | 1 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 1 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Mechanical ileus (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Autoimmune colitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 3
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2
Intussusception (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 1 | 3
Cardiac failure (Cardiac disorders) | 2 | 0 | 4
Pericardial effusion (Cardiac disorders) | 2 | 3 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1 | 1
Myocarditis (Cardiac disorders) | 1 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 0
Ventricle rupture (Cardiac disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 4
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Cardiac hypertrophy (Cardiac disorders) | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 2
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Toxic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Brachial plexopathy (Nervous system disorders) | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 1 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Coma (Nervous system disorders) | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Facial paralysis (Nervous system disorders) | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 1 | 2
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Myasthenic syndrome (Nervous system disorders) | 0 | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 3
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 2
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumor compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Superior vena cava syndrome (Vascular disorders) | 3 | 0 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 2 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 1
Peripheral ischemia (Vascular disorders) | 1 | 1 | 0
Shock hemorrhagic (Vascular disorders) | 1 | 1 | 1
Thrombosis (Vascular disorders) | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0
Arterial thrombosis (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Inferior vena caval occlusion (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 2 | 0
Blood sodium decreased (Investigations) | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0
Troponin T increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 2
Weight decreased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Dermatitis exfoliative generalized (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Haematotoxicity (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Myelosuppression (Blood and lymphatic system disorders) | 0 | 0 | 2
Hypothyroidism (Endocrine disorders) | 2 | 0 | 1
Goiter (Endocrine disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Immune-mediated hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Thyroiditis (Endocrine disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1
Hypopituitarism (Endocrine disorders) | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 3 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 3 | 0
Cholecystitis (Hepatobiliary disorders) | 3 | 0 | 1
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Breath holding (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 0
Nephritis (Renal and urinary disorders) | 1 | 0 | 0
Nephropathy (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 2 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Macular fibrosis (Eye disorders) | 1 | 0 | 0
Swelling of eyelid (Eye disorders) | 0 | 0 | 1
Aplasia (Congenital, familial and genetic disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab Biweekly (N=361) | Avelumab Weekly (N=318) | Chemotherapy (N=500)
Asthenia (General disorders) | 58 | 54 | 74
Fatigue (General disorders) | 58 | 56 | 99
Pyrexia (General disorders) | 51 | 50 | 32
Chills (General disorders) | 28 | 20 | 2
Non-cardiac chest pain (General disorders) | 15 | 12 | 16
Oedema peripheral (General disorders) | 14 | 9 | 48
Chest pain (General disorders) | 13 | 15 | 10
Influenza like illness (General disorders) | 10 | 1 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 50 | 50 | 49
Cough (Respiratory, thoracic and mediastinal disorders) | 48 | 41 | 45
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 25 | 23 | 23
Productive cough (Respiratory, thoracic and mediastinal disorders) | 14 | 8 | 14
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 11
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Weight decreased (Investigations) | 37 | 32 | 41
Alanine aminotransferase increased (Investigations) | 31 | 37 | 37
Aspartate aminotransferase increased (Investigations) | 24 | 22 | 30
Lipase increased (Investigations) | 20 | 17 | 11
Gamma-glutamyltransferase increased (Investigations) | 19 | 20 | 22
Blood creatinine increased (Investigations) | 16 | 12 | 30
Amylase increased (Investigations) | 15 | 17 | 17
Weight increased (Investigations) | 15 | 12 | 8
Blood creatine phosphokinase increased (Investigations) | 8 | 10 | 4
Platelet count decreased (Investigations) | 6 | 2 | 43
Blood lactate dehydrogenase increased (Investigations) | 5 | 3 | 4
Neutrophil count decreased (Investigations) | 2 | 2 | 62
Blood calcium decreased (Investigations) | 1 | 0 | 1
C-reactive protein increased (Investigations) | 1 | 6 | 4
White blood cell count decreased (Investigations) | 1 | 1 | 39
White blood cell count increased (Investigations) | 1 | 2 | 1
Constipation (Gastrointestinal disorders) | 59 | 21 | 87
Nausea (Gastrointestinal disorders) | 41 | 33 | 164
Diarrhoea (Gastrointestinal disorders) | 37 | 39 | 47
Vomiting (Gastrointestinal disorders) | 19 | 24 | 73
Dyspepsia (Gastrointestinal disorders) | 12 | 2 | 16
Dysphagia (Gastrointestinal disorders) | 5 | 6 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 1 | 7
Haemorrhoids (Gastrointestinal disorders) | 2 | 3 | 4
Odynophagia (Gastrointestinal disorders) | 1 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 25 | 21 | 21
Nasopharyngitis (Infections and infestations) | 23 | 11 | 16
Pneumonia (Infections and infestations) | 23 | 24 | 28
Respiratory tract infection (Infections and infestations) | 13 | 6 | 12
Bronchitis (Infections and infestations) | 12 | 9 | 12
Urinary tract infection (Infections and infestations) | 12 | 14 | 17
Decreased appetite (Metabolism and nutrition disorders) | 65 | 61 | 90
Hypoalbuminaemia (Metabolism and nutrition disorders) | 14 | 20 | 12
Hyponatraemia (Metabolism and nutrition disorders) | 12 | 16 | 15
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 10 | 21
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 5 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 50 | 31 | 31
Back pain (Musculoskeletal and connective tissue disorders) | 39 | 29 | 34
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 15 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 12 | 20
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 14 | 12 | 15
Bone pain (Musculoskeletal and connective tissue disorders) | 10 | 6 | 9
Flank pain (Musculoskeletal and connective tissue disorders) | 6 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 12
Rash (Skin and subcutaneous tissue disorders) | 30 | 27 | 36
Pruritus (Skin and subcutaneous tissue disorders) | 26 | 28 | 15
Dry skin (Skin and subcutaneous tissue disorders) | 19 | 12 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 3 | 30
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 3 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Headache (Nervous system disorders) | 24 | 21 | 24
Dizziness (Nervous system disorders) | 20 | 12 | 29
Hypoaesthesia (Nervous system disorders) | 5 | 2 | 5
Paraesthesia (Nervous system disorders) | 5 | 5 | 14
Taste disorder (Nervous system disorders) | 0 | 0 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 52 | 28 | 2
Anaemia (Blood and lymphatic system disorders) | 37 | 57 | 232
Leukopenia (Blood and lymphatic system disorders) | 6 | 2 | 42
Neutropenia (Blood and lymphatic system disorders) | 6 | 3 | 113
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 8 | 60
Leukocytosis (Blood and lymphatic system disorders) | 1 | 3 | 0
Hypertension (Vascular disorders) | 22 | 13 | 20
Hypotension (Vascular disorders) | 11 | 1 | 8
Hot flush (Vascular disorders) | 1 | 1 | 2
Insomnia (Psychiatric disorders) | 29 | 13 | 33
Depression (Psychiatric disorders) | 6 | 2 | 8
Confusional state (Psychiatric disorders) | 2 | 2 | 2
Hypothyroidism (Endocrine disorders) | 24 | 21 | 8
Atrial fibrillation (Cardiac disorders) | 10 | 4 | 3
Tachycardia (Cardiac disorders) | 5 | 9 | 7
Vision blurred (Eye disorders) | 3 | 0 | 2
Vitreous floaters (Eye disorders) | 1 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5 | 0
Contrast media allergy (Immune system disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT02576574/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT02576574/SAP_001.pdf